CLINICAL TRIAL: NCT02762552
Title: Micro-embolic Signals Detection With Transcranial HOLter in Acute Ischemic STroke: Yield in the Etiologic woR-kup
Brief Title: Micro-embolic Signals Detection With Transcranial HOLter in Acute Ischemic STroke
Acronym: HOLISTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/14
Record Dates: First submitted 2015-08-07; First posted 2016-05-05 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: Stroke; Etiology; Recurrence; Transcranial holter; Microembolic signals
MeSH Terms: conditions — Stroke; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial-holter monitoring (Experimental): Transcranial doppler in patient with ischemic stroke
  Interventions: Device: Transcranial-holter monitoring

INTERVENTIONS:
Device: Transcranial-holter monitoring — Transcranial holter with an 4 hour-recording

SUMMARY:
In acute ischemic stroke, the identification of an etiology is of major importance to prevent recurrence by providing the best treatment. Because of numerous possible underlying etiologies, the etiological work-up of ischemic stroke includes a wide range of diagnostic tests, which can be invasive, long and expensive. Moreover, many patients receive a diagnosis of undetermined stroke even after all available diagnosis tests are done, precluding optimal treatment.

DETAILED DESCRIPTION:
Asymptomatic MES detected by transcranial doppler have been reported in patient with ischemic stroke. It has been previously demonstrated that MES predict stroke recurrence and that the frequency of MES depends on stroke etiology. However, the pattern of MES has never been correlated to stroke etiology. Transcranial-holter is a novel ambulatory system which allows prolonged recording (up to 4 hours) leading to an increased detection of MES.

Therefore, transcranial holter with an 4 hour-recording will be performed for consecutive eligible patients hospitalized in our stroke care unit. During the recording, the patient will be able to continue their usual activities (eating, walking, speaking and sleeping).

All the included patients will have a classical follow-up at 3, 6 months and 12 months. The neurologist, blinded to the results of transcranial-holter, will have to prescribe and analyze the results of diagnostic tests to identify stroke etiology. Stroke etiology will be established according to the ASCOD classification. Questioning and neurological exam (NIHSS score) will be performed looking for potential recurrent stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke in the middle cerebral artery territory
* Acute ischemic stroke within the 7 first days from the onset of the symptoms
* Patient hospitalized in our stroke care unit
* Man or woman older than 18 years
* Patient affiliated to a social security system
* Free Consent, informed writing signed by the participant or the person of confidence and the investigator (no later than the day of inclusion and before any examination required by research)

Exclusion Criteria:

* Transient ischemic stroke
* Ischemic stroke in the vertebro-basilar or anterior cerebral artery territory.
* Proximal middle cerebral artery occlusion leading to the impossibility of recording
* Patient who could not express his consent
* Patient under guardianship or judicial protection
* Pregnant or breastfeeding woman
* Emergency situation
* Life expectancy under 6 months

Exclusion criteria (after inclusion) :

* Absent of bilateral Acoustic window
* Analyzable Recording <30min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Pattern of Microembolic signals (MES) recorded by Transcranial-holter monitoring and interpreted by an observer (index test) | Day 0 (inclusion)
  Microembolic signals (MES) will be recorded using Transcranial-holter monitoring (index test) for 4 hours at the acute phase of ischemic stroke. The pattern will be described (frequency, laterality) by the observer interpreting recordings, blinded to stroke etiology as established by the reference standard.
Etiology of ischemic stroke according to ASCOD phenotyping (A: atherosclerosis; S: small-vessel disease; C: cardiac pathology; O: other causes D: dissection) (reference standard) | Month 12
  Etiologic work-up of ischemic stroke will result in ASCOD classification (reference standard) of etiology. Work-up and classification will be established blind to the pattern of microembolic signals recordede by Transcranial-holter monitoring (index test)

SECONDARY OUTCOMES:
Stroke recurrence | Month 12
  Existence of a stroke recurrence will be assessed by clinical examination and possibly additional tests (imaging,..)
Actual duration of Transcranial-holter monitoring recording | Day 0 (inclusion)
  Actual duration of Transcranial-holter monitoring recording (minutes) will be measured (expected duration 4 hours) as a feasibility criterion

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Renou, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France